CLINICAL TRIAL: NCT03871712
Title: Return to Work for People With Musculoskeletal Disorders: A Randomized Controlled Trial of the Effectiveness of Usual Case Management Compared to Usual Case Management Plus Motivational Interviewing or Stratified Vocational Advice Intervention. The MI-NAV Study
Brief Title: Effectiveness of Motivational Interviewing on Return to Work in People on Sick Leave Due to Musculoskeletal Disorders
Acronym: MI-NAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Norwegian Labour and Welfare Administration (Other)
Responsible Party: Principal Investigator, Britt Elin Øiestad, Associate Professor, Oslo Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: The MI-NAV Study
Record Dates: First submitted 2019-02-27; First posted 2019-03-12 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Musculoskeletal Disease; Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Diseases; Musculoskeletal Pain | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: A multi-arm randomised controlled trial with two intervention groups and one control group doing as usual (ordinary NAV practice).
  The allocation will be prepared with block randomisation for risk of long term sick leave as predicted by the Orebro Screening Questionnaire and The Keele STarT MSK Tool. Preliminary data suggests a low/medium risk group (80% of the recruited participants) and a high risk group (20%). These numbers were calculated in another study of individuals on sick leave in Norway.
Who Masked: Investigator, Outcomes Assessor
Masking Description: In the written consent, the three groups will be described. Thus the participants will understand which group they are in after the first telephone call, and consequently not be blinded. The interventions are:
  1. Motivational interview by 2 meetings between participant and the NAV case-worker. Both the NAV case-workers and the participants will know that the intervention is motivational interviewing because it is only in this arm a NAV case-worker will do the intervention.
  2. Stratified vocational advice intervention (SVAI): a physiotherapist will call the study participants, and both the physiotherapist and the participants will know that they are in the SVAI intervention group from the informed consent.
  The researchers will be blinded to group allocation throughout the study recruitment and assessment up to the 6-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motivational Interview (MI) (Experimental): In the MI arm, a NAV case worker will meet the participants after the baseline assessment (electronic questionnaires) and randomisation and conduct the MI. The NAV case-worker will either meet (or call) again after a few weeks (anticipated 2-4 weeks) and conduct another MI.
  Interventions: Behavioral: Motivational interview
- Stratified vocational advice intervention (SVAI) (Active Comparator): A trained physiotherapist will call the participants after the baseline assessment and randomisation. The SVAI intervention will be stratified due to the participants risk of long term sick leave estimated by the Orebro Screening Questionnaire and The Keele STarT MSK Tool. The low/moderate risk group will receive 1-2 phone calls, and the high risk group will be followed up 2-4 times. The follow-up can include face to face Meetings bewteen the Physical therapist and the participant, and also the employer and general practitioner when needed. The intervention will include an assessment of the participants obstacles for returning to work and help to develop and implement an action plan to overcome obstacles. The physical therapists' will cooperate with other health care providers and employer when needed.
  Interventions: Behavioral: Stratified vocational advice
- Usual follow-up (No Intervention): This arm will be the control group receiving usual NAV follow-up. The other two groups will also receive usual NAV follow-up additionally to the interventions.

INTERVENTIONS:
Behavioral: Motivational interview — The participants will be called twice with 2-4 weeks interval after the randomisation. This will be after 8 weeks of sick leave.
  Arms: Motivational Interview (MI)
Behavioral: Stratified vocational advice — The participants will be called after the randomisation. The amount of calls/meetings will be decided after each call, but with a maximum of 4 for the high risk group. This may include physical meetings.
  Other Names: Vocational advice
  Arms: Stratified vocational advice intervention (SVAI)

SUMMARY:
Musculoskeletal disorders are the main causes for sickness absence and disability benefits in Norway and the leading causes of disability worldwide. There is strong evidence that long-term sickness absence due to musculoskeletal disorders provides a poor prognosis, both in terms of work-related disability, physical and mental health, and health related quality-of-life. To assist people return to work a range of vocational rehabilitation programs exist, but the initiatives have not been able to reduce the number of people who are on sick leave due to musculoskeletal disorders. In Norway, The Norwegian Labour and Welfare Administration (NAV) case-workers have taken such approaches in use, primarily by teaching their employees with user contact in how to use Motivational Interviewing (MI). However, the evidence on the effectiveness of MI on return to work is highly uncertain. The objectives of this project are to compare the effectiveness and cost-effectiveness of usual case management alone with usual case management plus MI or usual case management plus stratified vocational advice intervention (SVAI), on RTW among people on sick leave due to musculoskeletal (MSK) disorders. All musculoskeletal diagnoses will be included. A multi-arm randomised controlled trial with 150 participants in each group will be conducted within the NAV system in Norway to evaluate these research questions.

DETAILED DESCRIPTION:
The main objective of this project is to evaluate the effectiveness of usual case management plus motivational interviewing (MI), provided by trained Norwegian Labour and Welfare Administration (NAV) case-workers, and usual case management plus a Stratified Vocational Advice Intervention (SVAI), including principles of MI and vocational advice provided by trained physiotherapists, compared to usual case management alone on return to work among people on sick leave due to a musculoskeletal disorder. A multi-arm randomised controlled trial (RCT) will be conducted in order to respond to the following specific research questions:

RQ 1a Is there a difference between usual case management plus MI and usual case management alone in reducing sickness absence days at 6 months follow-up among individuals who have been on sick leave for >7 weeks due to a musculoskeletal disorder?

RQ 1b Is there a difference between usual case management plus SVAI and usual case management alone in reducing sickness absence days at 6 months follow-up among individuals who have been on sick leave for >7 weeks due to a musculoskeletal disorder?

RQ 2a Is there a difference between usual case management plus MI and usual case management alone in reducing sickness absence days at 12 months follow-up among individuals who have been on sick leave for >7 weeks due to a musculoskeletal disorder?

RQ 2b Is there a difference between usual case management plus SVAI and usual case management alone in reducing sickness absence days at 12 months follow-up among individuals who have been on sick leave for >7 weeks due to a musculoskeletal disorder?

RQ 3a Is there a difference between usual case management plus MI and usual case management alone in time until sustained RTW during 12 months follow-up among individuals who have been on sick leave for >7 weeks due to a musculoskeletal disorder?

RQ 3b Is there a difference between usual case management plus SVAI and usual case management alone in time until sustained RTW during 12 months of follow-up among individuals who have been on sick leave for >7 weeks due to a musculoskeletal disorder?

RQ 4a Is there a difference in the proportions of participants who receive sick leave benefits each month during 12 months of follow-up between usual case management plus MI compared to usual case management alone?

RQ 4b Is there a difference in the proportion of individuals who receive sick leave benefits each month during 12 months of follow-up between usual case management plus SVAI compared to usual case management alone?

RQ 5a Is there a difference in cost-effectiveness, cost-utility and cost-benefit during 6 months of follow-up between individuals on sick leave with musculoskeletal disorders who receive usual case management plus MI compared to those who receive usual case management alone?

RQ 5b Is there a difference in cost-effectiveness, cost-utility and cost-benefit during 6 months of follow-up between individuals on sick leave with musculoskeletal disorders who receive usual case management plus SVAI compared to those who receive usual case management alone?

RQ 6a Is there a difference in cost-effectiveness, cost-utility and cost-benefit during 12 months of follow-up between individuals on sick leave with musculoskeletal disorders who receive usual case management plus MI compared to those who receive usual case management alone?

RQ 6b Is there a difference in cost-effectiveness, cost-utility and cost-benefit during 12 months of follow-up between individuals on sick leave with musculoskeletal disorders who receive usual case management plus SVAI compared to those who receive usual case management alone?

RQ 7a Is there a difference in musculoskeletal health during 12 months of follow up between individuals on sick leave with musculoskeletal disorders who receive usual case management plus MI compared to those who receive usual case management alone?

RQ 7b Is there a difference in musculoskeletal health during 12 months of follow up between individuals on sick leave with musculoskeletal disorders who receive usual case management plus SVAI compared to those who receive usual case management alone?

The following hypotheses will be tested:

H 1a There is no difference in number of sickness absence days between participants who receive usual case management plus MI compared to those who receive usual case management alone at 6 months follow-up.

H 1b There is no difference in number of sickness absence days between participants who receive usual case management plus SVAI compared to those who receive usual case management alone at 6 months follow-up.

H 2a There is no difference in number of sickness absence days between participants who receive usual case management plus MI compared to those who receive usual case management alone at 12 months follow-up.

H 2b There is no difference in number of sickness absence days between participants who receive usual case management plus SVAI compared to those who receive usual case management alone at 12 months follow-up.

H 3a There is no difference in time until first sustained RTW between participants who receive usual case management plus MI compared to those who receive usual case management alone during 12 months follow-up.

H 3b There is no difference in time until first sustained RTW between participants who receive usual case management plus SVAI compared to those who receive usual case management alone during 12 months of follow-up.

H 4a There is no difference in the proportions of participants who receive sick leave benefits each month between usual case management plus MI compared to usual case management alone during 12 months of follow-up.

H 4b There is no difference in the proportions of individuals receiving sick leave benefits each month between usual case management plus SVAI compared to usual case management alone during 12 months of follow-up.

H 5a There is no difference in cost-effectiveness, cost-utility and cost-benefit between usual case management plus MI compared to usual case management alone during 6 months of follow up.

H 5b There is no difference in cost-effectiveness, cost-utility and cost-benefit between usual case management plus SVAI compared to usual case management alone during 6 months of follow up.

H 6a There is no difference in cost-effectiveness, cost-utility and cost-benefit between usual case management plus MI compared to usual case management alone during 12 months of follow up.

H 6b There is no difference in cost-effectiveness, cost-utility and cost-benefit between usual case management plus SVAI compared to usual case management alone during 12 months of follow up.

H 7a There is no difference in musculoskeletal health between participants who receive usual case management plus MI compared to those who receive usual case management alone during 12 months of follow-up.

H 7b There is no difference in musculoskeletal health between participants who receive usual case management plus SVAI compared to those who receive usual case management alone during 12 months of follow-up.

A multi-arm RCT with a full-scale health economic evaluation and mediator analysis will be conducted. In order to avoid contextual contamination effect only NAV offices in which the employees have not received any previous MI training will be included. All eligible participants will be asked to participate.

The head NAV office in Oslo will provide weely lists of persons meeting the eligibility criteria. We will contact eligible people by phone and give information about the study. Elibible persons who are interested will then receive a link to the informed consent and the baseline questionnaire.

MI intervention: In addition to usual case management, the MI group will receive 2 motivational interviews provided by a NAV case-worker. The case-workers will be educated and mentored throughout the study period. The first MI will be face-to-face, while the second may by phone, but preferable face-to-face.The interviews will be given in week 8/9 of the sick leave period, and then again after approximately 2 weeks.

SVAI intervention: In addition to usual case management, the SVAI group will be followed up by trained physical therapists. This group will be stratified into risk groups for long term sick leave; an "at risk group" and a "high risk group". The at risk group will receive 1-2 phone calls with emphasis on identifying obstacles for return to work, and solutions for resolving these obstacles. The high risk group will be followed up 3-4 times. The first follow-up is by phone, the remaining follow-ups can be either by phone or face to face meetings and can include a workplace visit. The SVAI intervention will end before week 26 of the participants' sick leave period.

Usual case management: The Norwegian welfare state has a system for following up people on sick leave, including a follow-up plan developed by the worker and the employer by week 4 of the sick leave period, a dialogue meeting between the worker and the employer by week 7, and a second dialogue Meeting including a NAV caseworker, by week 26.

The study flow:

Baseline recruitment will occur by week 8 of the sick leave period. The two interventions will start immediately after randomization and baseline assessments. The questionnaires will be sent electronic through a secure system from University of Oslo at baseline, and after 3, 6, 9, and 12 months.

A pilot study will be conducted prior to start of the RCT to test the study protocol including the recruitment procedure, the randomisation procedure, the information flow between researchers, physical therapists, NAV case workers and study participants, and the interventions (MI and SVAI). The pilot study will end by the first 100 included participants (August 31. 2019). The participants in the pilot study will be included in the RCT as long as the protocol will not be changed with respect to the scientific method and research questions (internal pilot study).

A fidelity study of the MI and SVAI interventions will be conducted to measure how well the trained personnel is using the methods and interventions as intended. For the MI arm, a developed instrument (Motivational Interviewing Treatment Integrity Coding Manual 4.2.1) will be used to score the feasibility from audio recordings of all NAV case-workers who do the MI intervention. For the SVAI intervention, feasibility will be measured by both audiotaping and from the telephone script/journal that the SVAI physiotherapists fill out during the talk with the study participant. The investigators plan to do 20-25 audiotapes of the 5 SVAI physiotherapists.

ELIGIBILITY:
Inclusion Criteria:

* Have musculoskeletal disorders
* Live in South-East Norway
* Have been on sick leave for 8 weeks with a current sick-leave status of 50%-100%
* Have a job to return to

Exclusion Criteria:

* Have serious somatic or psychological disorders (e.g. cancer, psychotic disorders)
* Have specific disorder requiring specialized, ongoing treatment;
* Are pregnant
* Are self-employed or work free lance
* Have insufficient Norwegian or English speaking or writing skills to participate in group session and fill out questionnaire.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Sickness absence days | 6 months
  Total number of sickness absence days up to the 6-month's follow-up

SECONDARY OUTCOMES:
Sickness absence days | 12 months
  Total number of sickness absence days up to the 12-month's follow-up
Sustainable return to work | 12 months
  Time in months until full sustainable return to work during 12 months of follow-up, defined as 4 weeks of 100% return to original employment fraction without relapse, obtained from national registers.
Medical benefits | 12 months
  The chance of receiving medical benefits during 12 months of follow-up measured as repeated events assessed with data from national registers.
Cost-utility | 6 months
  Cost-utility at 6 months assessed by healthcare utilisation obtained from national registries. To measure treatment effects and health utilities the Euro Quality of Life 5 Dimentions 5 Levels (EQ-5D-5L) utility index will be used. The EQ-5D-5L is a generic and preference-weighted measure of health-related quality-of-life based on five dimensions: mobility, self-care, activities of daily life, pain, and anxiety and/or depression. For each dimension, the patient assesses five possible levels of problems (from no to severe, 1-5). Health gains will be expressed as quality-adjusted life years (QALYs), which will be derived from the EQ-5D-5L utility scores, using the UK tariff. QALYs range from -0.59 to 1, where 1 corresponds to perfect health, and -0.59 to worst imaginable health.
Cost-utility | 12 months
  Cost-utility at 12 months assessed by healthcare utilisation obtained from national registries. To measure treatment effects and health utilities the Euro Quality of Life 5 Dimentions 5 Levels (EQ-5D-5L) utility index will be used. The EQ-5D-5L is a generic and preference-weighted measure of health-related quality-of-life based on five dimensions: mobility, self-care, activities of daily life, pain, and anxiety and/or depression. For each dimension, the patient assesses five possible levels of problems (from no to severe, 1-5). Health gains will be expressed as quality-adjusted life years (QALYs), which will be derived from the EQ-5D-5L utility scores, using the UK tariff. QALYs range from -0.59 to 1, where 1 corresponds to perfect health, and -0.59 to worst imaginable health.
Cost-effectiveness | 6 months
  Cost-effectiveness at 6 months assessed by healthcare utilisation obtained from national registries.
Cost-effectiveness | 12 months
  Cost-effectiveness at 12 months assessed by healthcare utilisation obtained from national registries.
Musculoskeletal health | 12 months
  Musculoskeletal health will be assessed at the 12 month's follow-up with the Musculoskeletal Health Questionnaire (MSK-HQ). MSK-HQ is a new outcome questionnaire with 14 items capturing a broad variety of musculoskeletal conditions. The score provides a range from 0 to 56, with higher scores indicating better MSK health status.The MSK-HQ has undergone initial psychometric testing in four different musculoskeletal cohorts and demonstrated high completion rates, excellent test-retest reliability and strong convergent validity with other disease-specific outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Hege Bentzen, PhD, Study Director — OsloMet - Oslo Metropolitan University
Locations (1):
- Oslo Metropolitan Universtiy, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Killingmo RM, Rysstad T, Maas E, Pripp AH, Aanesen F, Tingulstad A, Tveter AT, Oiestad BE, Grotle M. Modifiable prognostic factors of high societal costs among people on sick leave due to musculoskeletal disorders: a replication study. BMC Musculoskelet Disord. 2024 Dec 3;25(1):990. doi: 10.1186/s12891-024-08132-3. PMID 39627785
- [Derived] Tingulstad A, Maas ET, Rysstad T, Oiestad BE, Aanesen F, Pripp AH, Van Tulder MW, Grotle M. Six-month cost-effectiveness of adding motivational interviewing or a stratified vocational advice intervention to usual case management for workers with musculoskeletal disorders: the MI-NAV economic evaluation. J Occup Med Toxicol. 2023 Nov 14;18(1):25. doi: 10.1186/s12995-023-00394-2. PMID 37964240
- [Derived] Cashin AG, Oiestad BE, Aanesen F, Storheim K, Tingulstad A, Rysstad TL, Lee H, McAuley JH, Sowden G, Wynne-Jones G, Tveter AT, Grotle M. Mechanisms of vocational interventions for return to work from musculoskeletal conditions: a mediation analysis of the MI-NAV trial. Occup Environ Med. 2023 May;80(5):246-253. doi: 10.1136/oemed-2022-108716. Epub 2023 Mar 2. PMID 36863864
- [Derived] Aanesen F, Grotle M, Rysstad TL, Tveter AT, Tingulstad A, Lochting I, Smastuen MC, van Tulder MW, Berg R, Foster NE, Wynne-Jones G, Sowden G, Fors E, Bagoien G, Hagen R, Storheim K, Oiestad BE. Effectiveness of adding motivational interviewing or a stratified vocational advice intervention to usual case management on return to work for people with musculoskeletal disorders: the MI-NAV randomised controlled trial. Occup Environ Med. 2023 Jan;80(1):42-50. doi: 10.1136/oemed-2022-108637. Epub 2022 Nov 25. PMID 36428098
- [Derived] Oiestad BE, Aanesen F, Lochting I, Storheim K, Tingulstad A, Rysstad TL, Smastuen MC, Tveter AT, Sowden G, Wynne-Jones G, Fors EA, van Tulder M, Berg RC, Foster NE, Grotle M. Study protocol for a randomized controlled trial of the effectiveness of adding motivational interviewing or stratified vocational advice intervention to usual case management on return to work for people with musculoskeletal disorders. The MI-NAV study. BMC Musculoskelet Disord. 2020 Jul 28;21(1):496. doi: 10.1186/s12891-020-03475-z. PMID 32723318

DOCUMENTS (3):
  • Statistical Analysis Plan: Effectiveness of MI and SVAI on sick leave (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT03871712/SAP_000.pdf
  • Statistical Analysis Plan: Moderation analysis of MI and SVAI on sick leave (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT03871712/SAP_001.pdf
  • Statistical Analysis Plan: Modifiable prognostic factors of high costs (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT03871712/SAP_002.pdf